CLINICAL TRIAL: NCT06260371
Title: National Observatory of Mycoplasma Infections in Hospitalized Children Under 18 Ages in France
Brief Title: National Observatory of Mycoplasma Infections in Children Under 18 Ages in France
Acronym: ORIGAMI
Status: Recruiting | Type: Observational
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Collaborators: Groupe de Pathologies Infectieuses Pédiatriques (GPIP) (Other)
Responsible Party: Sponsor
Other Study IDs: ORIGAMI
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-01

CONDITIONS: Mycoplasma Infections; Hospitalized Children
MeSH Terms: conditions — Mycoplasma Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — nasopharyngeal, oropharyngeal, lung, pleural puncture, pleural fluid, skin swab, cerebrospinal fluid, biopsy, etc... taken during routine care may be stored at hospital and analysed later. These data could be explored during end-of-study analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was set up because of an unusual increase in the number of cases of mycoplasma infections in France between June and November 2023.

Clinical data from children with mycoplasma infections will be collected to characterise this infection and facilitate hospital management.

DETAILED DESCRIPTION:
In this study, the number of cases will be collected. In addition, we will determine the clinical, biological and microbiological characteristics of these cases.

These following data will be collected: signs or symptoms associated with this infection, clinical complications, biological and microbiological tests done during hospitalisation, treatment used during hospitalization, results of thoracic x-ray and lung ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years (only hospitalized children)
* Documented mycoplasma infection (positive multiplex PCR and/or positive serology)

Exclusion Criteria:

* Refusal by one of the parents or by Child in understanding age

Ages: 1 Day to 17 Years | Sex: All
Age Groups: Child
Study Population: hospitalised children under 18 age, with Mycoplasma infection
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients hospitalized for mycoplasma infections | 1 year
  Proportion of hospitalized children due to mycoplasma infections
medical characterisation of mycoplasma infections | 1 year
  Assessment of clinical, biological and microbiological characteristics of mycoplasma infections cases.

SECONDARY OUTCOMES:
Identify risk factors of serious infection | 1 year
  Describe what is responsible of serious infection.
Identify predictive signs of serious infection | 1 year
  what are the warning signs of a serious infection?
Type of complications | 1 year
  Describe any complications due to infection
Patients outcome | 1 year
  Proportion of patients recovered
healthcare used for infected children | 1 year
  Describe healthcare provided during hospitalisation of infected children in order to manage this type of infection
treatment used during hospitalisation | 1 year
  type of treatment used during hospitalisation to manage the infection
clinical description of infected children | 1 year
  clinical description of all cases of mycoplasma infections reported during the study
Type of mycoplasma involved in infected children | 1 year
  characterisation of mycoplasma involved in infection (strain, molecular epidemiology and antibiotic resistance)
performance of complementary diagnostic tests for lung disorders | 1 year
  for lung disorders, assessment of performance of complementary diagnostic tests (chest X-ray, lung ultrasound, C reactive protein (CRP), multiplex polymerase chain reaction (PCR), etc).
compare medical data collected during hospitalisation | 1 year
  Assessment of the correlation between clinical, radiological and biological data of infected children

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Levy, Study Director — Association Clinique Thérapeutique Infantile du val de Marne; Anais Chosidow, Principal Investigator — Hôpital Intercommunal de Villeneuve-Saint-Georges; Emilie Pauquet, Principal Investigator — Hôpital des Enfants, CHU de Bordeaux
Locations (1):
- ACTIV, Créteil, France

REFERENCES:
- [Derived] Chosidow A, Maakaroun-Vermesse Z, Ok V, Delecroix C, Le Roux P, Dommergues MA, de Larminat J, Jeziorski E, Ronjat P, Jaume L, Welfringer-Morin A, Bebear C, Gits-Muselli M, Viriot D, Roux CJ, Bechet S, Romain AS, Lorrot M, Cohen R, Levy C, Cohen JF; ORIGAMI Study Group. Post-COVID-19 resurgence of Mycoplasma pneumoniae infections in French children (ORIGAMI): a retrospective and prospective multicentre cohort study. Lancet Infect Dis. 2025 Nov 19:S1473-3099(25)00598-5. doi: 10.1016/S1473-3099(25)00598-5. Online ahead of print. PMID 41274297